CLINICAL TRIAL: NCT05303571
Title: Project Bidof - Achieving Hybrid Monovision by Pairing Bifocal and EDOF Lens Technology
Brief Title: Project Bidof - Monovision by Pairing Bifocal and EDOF Lens
Acronym: Bidof
Status: Withdrawn | Type: Observational
Why Stopped: not feasible
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Principal Investigator, Matthias Bolz, Head of Ophtalmology, Johannes Kepler University of Linz
Other Study IDs: KUK-Ophthalmology-005
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Monodof: monofocal and EDOF lens
- Bidof: Bifocal and EDOF lens

SUMMARY:
Modern day cataract surgery isn't just a rehabilitative procedure anymore but rather aims at improving a patient's quality of life by reducing the need for spectacles in everyday life to a minimum. One way of achieving this goal is by using different lens technologies, such as a mono- or bifocal lens paired a lens with EDOF technology, as EDOF lenses provide an enhanced depth of focus by creating a single elongated focal point. As this method is well established, the aim of this study is to compare the monofocal/EDOF cohort to the bifocal/EDOF cohort and evaluate visual acuity and patient satisfaction for both combinations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 99 years
* signed informed consent form
* condition after cataract surgery

Exclusion Criteria:

* no signed informed consent form
* laser treatment of the Cornea
* macular pathologies
* corneal pathologies
* irregular astigmatism
* pregnancy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient between 21 and 99 years after cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Distance Visual Acuity | 6 months
  percentage of patients with binocular distance corrected visual acuity of logMAR > 0.2
Intermediate Visual Acuity | 6 months
  percentage of patients with binocular intermediate distance corrected visual acuity of logMAR > 0.2
Near Visual Acuity | 6 months
  percentage of patients with binocular near visual acuity logmar < 0.2

SECONDARY OUTCOMES:
contrast vision | 3 months
  contrast sensitivity vision
Halo and Glare | 3 months
  Halo and Glare Simulator
Defocus curve | 3 and 6 months
  Defocus curve

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Kepler University, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No